CLINICAL TRIAL: NCT03359447
Title: Effectiveness of Weekly and Daily Iron Supplementation for the Prevention of Iron-deficiency Anemia in Infants. Impact on Genomic Stability
Brief Title: Iron Deficiency Anemia, Iron Supplementation and Genomic Stability in Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20070773
Record Dates: First submitted 2017-11-13; First posted 2017-12-02 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Anemia; Iron-deficiency
Keywords: infant; primary prevention
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Two main arms: weekly vs daily iron supplementation. Infants who are exclusively breast fed will be randomized into three groups: no iron supplementation, weekly iron supplementation and daily iron supplementation. Infants that are partially fed with infant formula will be randomized into two groups: weekly iron supplementation and daily iron supplementation.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessor: the outcomes are defined by hemoglobin and ferritin (corrected by CRP), also genomic instability is defined by a laboratory result such as comet assay. The members of the laboratory will receive labeled specimens with a code unrelated to the allocated arm.
  The investigators that will analyze the data will not carry out the study. All the clinical data will be obtained by the care providers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Iron (Experimental): Weekly ferrous sulfate: one dose (4mg/kg/week).
  Interventions: Drug: Weekly Ferrous Sulfate
- Daily Iron (Active Comparator): Daily ferrous sulfate: one dose (1 mg/kg/day). Maximum daily dose: 40 mg
  Interventions: Drug: Daily Ferrous Sulfate

INTERVENTIONS:
Drug: Weekly Ferrous Sulfate — Drops
  Other Names: Fer-in-sol
  Arms: Weekly Iron
Drug: Daily Ferrous Sulfate — Drops
  Other Names: Fer-in-sol
  Arms: Daily Iron

SUMMARY:
This study compares weekly versus daily administration of iron for prevention of anemia in 6 months old infants. One third of the infants that are exclusively breast fed will not receive iron, the second third will receive iron weekly and the last third will receive iron daily. Half of the infants that take infant formula will receive iron weekly and the other half will receive iron daily.

DETAILED DESCRIPTION:
Iron deficiency is the most prevalent nutritional deficiency and the main cause of anemia. It's estimated that 43% of pre-school children worldwide are anemic, in Argentina a national survey carried out in 2007 (last survey), showed that 34.5% of children less than 2 years old were anemic and that 50.8% of children 6 to 9 months old were anemic. Although there is a consensus on iron supplementation as a preventive strategy for anemia in infants, there is a poor adherence due mainly to mild gastrointestinal adverse effects and low prescription rates from pediatricians. On the other hand, the excess of iron can lead to genomic instability with structural and functional alterations on proteins, lipids and DNA. Weekly administration of iron has been proposed as an alternative of similar efficacy and higher effectiveness in older children and pregnant women, but sufficient evidence for infants is lacking.

ELIGIBILITY:
Inclusion Criteria:

* 3 months old infants, clinically healthy, born to term (>37 weeks), that weighted at birth between 2500 and 4000 g, that have normal prenatal records.

Exclusion Criteria:

* anemic or iron deficient infants, or that have a chronic pathology, or that have undergone an acute pathology in the previous 15 days. Children that are receiving antibiotics or vitamin supplements.

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 204 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Anemia | 7 days
  Hemoglobin <11.0 g/dL in 6 months old infants.

SECONDARY OUTCOMES:
Iron deficiency | 7 days
  Serum Ferritin <12 ng/ml in 6 months old infants. If C-reactive protein > 5 mg/L, Iron deficiency is redefined as Serum Ferritin <30 ng/ml.
Adverse effects | Through study completion, an average of 1 year
  Frequency of at least one of the following during the three months intervention: rejection of food intake, constipation, vomiting, diarrhea, abdominal pain.
Genomic Instability | 15 days
  One of the following indicators is altered. Genomic damage: Comet assay: damage index (ID) over 200 cells. 8-oxo-dGuanosine.
  Oxidative Stress: catalase activity, superoxide dismutase activity, Tbars.
Adherence | Through study completion, an average of 1 year
  Low adherence: 1. Less than 50% of the drug was given to the infant (according to the remaining volume of the drug in its recipient) 2. Less tha 50% of the allocated intakes (according to care-taker registration on an almanaq)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Varea, Biochemist, Study Director — Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri
Locations (1):
- Instituto de Desarrollo e Investigaciones Pediátricas Prof. Dr. Fernando E. Viteri, La Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months following article publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.Proposals should be directed to enriqueflmartins@gmail.com To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (2):
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03359447/Prot_000.pdf
  • Informed Consent Form (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT03359447/ICF_001.pdf